CLINICAL TRIAL: NCT03272867
Title: Cross-over Randomized Placebo-controlled Pilot Study to Determine the Effect in Healthy Elderly Volunteers of the Anti-ageing Supplement "Promanna™" on a Number of Biomarkers Associated With DNA-damage and Oxidative Stress (PromAge)
Brief Title: Effect of an Anti-ageing Supplement on Oxidative Stress
Acronym: PromAge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Prof. dr. S.J.L. Bakker, MD, PhD, Prof. dr., University Medical Center Groningen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 14TGO01
Record Dates: First submitted 2017-09-02; First posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Healthy Volunteers; Age Group: 60-70; Overweight
MeSH Terms: conditions — Overweight | interventions — Proline; Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): One group of volunteers will ingest a powder with dose of 6.1 g ProManna twice a day for a period of 2 weeks
  Interventions: Dietary Supplement: ProManna
- Control group (Placebo Comparator): Another group of volunteers will ingest a powder with the same amount of a placebo twice a day for a periode of 2 weeks
  Interventions: Dietary Supplement: ProManna

INTERVENTIONS:
Dietary Supplement: ProManna
  Other Names: L-proline; D-mannitol

SUMMARY:
This pilot study serves to investigate whether ProManna intake leads to any changes in baseline levels for oxidative stress markers. In addition, biomarker responses following oxidative stress challenge tests will be assessed in subjects taking ProManna versus placebo supplements.

DETAILED DESCRIPTION:
Ageing is characterized by a progressive decline in the efficiency of physiological function and by the increased susceptibility to disease and death. Most ageing-associated diseases develop silently for many years before symptoms appear, leading to irreversible pathological conditions. Examples of these diseases are Alzheimer's, Parkinson's, osteoporosis, diabetes, cardiovascular disease and also cancer. Typically, patients are treated when most of the damage has already occurred, and existing drugs can rarely cure these diseases, but merely slow down further progression of the disease. Therefore, preventive measures that may delay the onset of these diseases can hold the best promise for healthy ageing. of the most plausible and acceptable explanations for the mechanistic basis of aging is the "free radical theory of aging". This theory postulates that aging and its related diseases are the consequence of free radical-induced damage to cellular macromolecules and the inability to counterbalance these changes by endogenous anti-oxidant defences. ProManna is a novel and safe food supplement that aims to decrease free radical-induced damage, thereby contributing to healthy ageing.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteer aged ≥ 60 to ≤ 70
2. Not involved in intensive sportive activities more than twice a week (e.g. playing football, tennis, running, cycling-racing, swimming)
3. Stable weight and no intention to lose weight until completion of the study (three times a day: a normal eating pattern).
4. Two weeks before the start and during the study no use of over the counter medication, prescribed medication, herbal medication or dietary supplements which in the investigator's opinion could affect study results, or which could be affected by the study product (i.e. absorption of oral medication will be influenced by D-Mannitol). Exception for sporadic use of paracetamol and/or treating an AE.
5. Able and motivated to comply with protocol requirements like for instance take the investigational product the way it is prescribed and to do the tests.
6. Voluntary signed written informed consent form (ICF) before the start of the pilot.

Exclusion Criteria:

1. BMI < 25 or > 30 kg/m2
2. Not being able to fast overnight (12 hours)
3. Diabetes mellitus
4. Gastrointestinal disorders
5. Undergone digestive tract surgery (except appendectomy)
6. Clinically significant inflammatory disease (possibly interfering with measurement of parameters in this study)
7. Weed smoking
8. Donation of blood within the last 3 months prior to admission to the clinic
9. Participation to another clinical study within 90 days before enrolment
10. Clinically relevant abnormalities in clinical chemistry or positive HIV, HbsAg and/or HepC at screening
11. Positive drug screen or alcohol breath test at D-1

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Changes in oxidative stress markers | Two weeks
Changes in oxidative stress following a hyperoxia or glucose challenge | Two weeks

SECONDARY OUTCOMES:
Changes in experienced health | Two weeks
  Rand-36-item Health Survey (SF-36)

CONTACTS AND LOCATIONS:
Locations (1):
- UMCG, Groningen, Netherlands